CLINICAL TRIAL: NCT03682341
Title: Study of the Relationship Between Oxidative Stress Gene Polymorphism and Individual Variation of Ovarian Reserve Function in Patients With Ovarian Endometrioma
Brief Title: Oxidative Stress Gene Polymorphism and Ovarian Reserve Functione
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: endometriosis oxidative stress
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Recruitment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients with ovarian endometriosis cyst
  Interventions: Genetic: endometriosis
- Group B: Patients with ovarian teratoma cyst
  Interventions: Genetic: endometriosis

INTERVENTIONS:
Genetic: endometriosis — patients with or without ovarian endometriosis

SUMMARY:
the relationship between FOXO3A-bim pathway gene polymorphisms and ovarian reserve function of paitients with ovarian endometrioma

DETAILED DESCRIPTION:
Ovarian reserve refers to the left ovarian cortex follicle growth, development, the quantity and quality of potential ability of oocytes, reflects the fertility in women. Ovarian endometrioms have an effect on ovarian reserve function. Oxidative stress is one of the important reasons. The effect has individual differences and the mechanisms are not clear.FOXO3A-bim pathway gene polymorphisms have been reported to related to individual variation of ovarian reserve function of paitients with POF. Our working hypothesis is that FOXO3A-bim pathway gene polymorphisms are also related to ovarian reserve function of paitients with ovarian endometrioma. In recent 10 years, we have set up a database including more than 2000 cases of ovarian endometrioma. In this project, we are going to investigate the oxidative stress factors, the level of sexual hormone, ultrasound information and the relationship between FOXO3A-bim pathway gene polymorphism.All these multi-diciplinary research will lead to novel understanding of individual variation of ovarian reserve function.

ELIGIBILITY:
Inclusion Criteria:

20 to 35 years old, non-menstrual period, not in pregnancy or puerperal period, diagnosed with ovarian cyst according to preoperative clinical symptoms, physical examination, ultrasound, CA125 and other non-surgical diagnosis methods, and all the participants having surgical indications, and ultimately conformed through histopathological diagnosis

Exclusion Criteria:

Participants receiving hormone therapy within the past six months, HIV or hepatitis B/C positive, autoimmune diseases, endocrine diseases and systemic diseases (such as diabetes, hormone therapy diseases, severe liver and kidney dysfunction), severe mental illness and malignant tumors.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with ovarian endometriosis cyst and teratoma cyst
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09-20 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
difference in ovarian reserve function | 4 months
  different ovarian reserve function in patients with or without ovarian endometriosis

SECONDARY OUTCOMES:
FOXO3A-bim pathway gene polymorphism | 4 months
  FOXO3A-bim pathway gene polymorphism in patients with or without ovarian endometriosis

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Leng, professor, Study Director — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li XY, Wang X, Gu ZY, Sun TT, Leng JH, Yu Q. Combined proteomics and transcriptomics identifies serpin family C member 1 associated protein as a biomarker of endometriosis. Ann Med. 2023;55(2):2243825. doi: 10.1080/07853890.2023.2243825. PMID 37572646